CLINICAL TRIAL: NCT04053166
Title: Effect of an Individualized Home-based Physical Activity Trial on Carotid Plaque Vulnerability for Asymptomatic Patients
Brief Title: Individualized Physical Activity and Carotid Plaque Instability
Acronym: PACAPh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 69HCL19_0345; 2019-A01543-54 (Other: ID-RCB)
Record Dates: First submitted 2019-08-06; First posted 2019-08-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Carotid Atherosclerosis
Keywords: Intraplaque haemorrhage; MRI; home-based Physical activity; carotic plaque vulnerability
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two experienced observers will blindly read the MRI scans.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized home-based physical activity (Experimental): The subjects of this arm will have a daily goal in number of steps based on the initial 2 first week evaluation of daily number of steps. They will wear connected wrists, and will be contacted twice a month by phone call by the adapted physical activity trainer to revaluate these goals.
  Interventions: Device: individualized home-based physical activity; Other: MRI; Biological: blood sampling; Other: Questionnaires; Other: 6-minute walk test
- Control group (Active Comparator): The subjects of this arm will not have evaluation of daily steps and recommendations regarding physical activity and sedentary behaviour. They will be asked to live as usual.
  Interventions: Other: MRI; Biological: blood sampling; Other: Questionnaires; Other: 6-minute walk test

INTERVENTIONS:
Device: individualized home-based physical activity — Subjects will have to reach a daily goal in number of steps, based on the initial evaluation, during 6 months . They will wear connected wrists, and will be contacted twice a month by phone call by an adapted physical activity to revaluate these goals.
  Arms: Individualized home-based physical activity
Other: MRI — An MRI will be performed for each patient at the end of the study to identify IPH and other features of histological vulnerability (lipid core, fibrous cap integrity and calcifications).
Biological: blood sampling — Blood will be collected, to analyse monocyte phenotype by flow cytometry, blood rheology by ektacytometry, coagulation by rotational thromboelastometry (ROTEM). Plasma will be extracted from blood to assess inflammation, oxidative stress and antioxidant markers.
Other: Questionnaires — sedentary, physical activity, nutrition and quality of life questionnaire will be performed fo each patient.
Other: 6-minute walk test — The 6-minute walk test is a simple, individualized test that measures how fast a patient walks on a flat, hard surface for 6 minutes.

SUMMARY:
Intraplaque hemorrhage (IPH) is one of the main features of the carotid plaque instability's and predictor of ischemic stroke. Benefits (on the basis on benefit/risk ratio) of the carotid endarterectomy remain unclear for stroke asymptomatic patients; thus, more and more patients with important stenosis (i.e. over 60%) detected are not operated. However, these patients need adapted therapeutic treatments to limit plaque instability and this should include physical activity (PA). Indeed, PA has been showed to decrease numerous inflammatory markers involved in atherosclerosis. It has also recently been reported on stroke asymptomatic patients that the prevalence of carotid IPH was decreased in those with higher level of PA. Magnetic Resonance Imaging (MRI) of the IPH has been shown to be the better non-invasive imaging technique to assess carotid plaque instability and in particular IPH. Here, the aim of this study is to assess the effect of an individualized home-based 6 months physical activity intervention on carotid IPH and other biomarkers of vulnerability for asymptomatic patients.

This study has been designed as a monocentric, longitudinal and interventional study. This study will involve one centre: Hopital Louis Pradel (HCL, Lyon). After inclusion tests, patients will be randomly included in the control group, or in the PA group. Patients of the PA group will have connected bracelets to measure daily count of steps. Twice a month, daily goals will be revaluated to increase or maintain the steps per day. The final goal is to reach 6 000 steps per day or increase by 30% the initial count of steps per day. Same tests will be done after 6 months of intervention for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an carotid atheromatous plaque with ≥ 50% North American Symptomatic Carotid Endarterectomy Trial (NASCET) stenosis
* Patient from vascular surgery department of the Louis Pradel Hospital of the Hospices Civils de Lyon, but not operated
* Males and females aged over 18 years old
* No contra-indication to physical activity with index performance (PS) < 2
* Available and voluntary to invest in the study throughout its duration (6 months)
* Able to understand, read and write French;
* a social security system or similar;
* Having dated and signed informed consent.

Exclusion Criteria:

* Transient ischemic attack (TIA) or ipsilateral cerebral infarction less than 6 months
* History of ipsilateral carotid surgery or cervical irradiation;
* Cancer, heart failure, seropositivity;
* Coronary risk;
* Renal failure (Cockcroft clearance of creatinine < 30 milliliter/minute (mL/min);
* Contraindication and precautions for use related to Prohance: hypersensitivity to the active substance or to any of the constituents of Prohance, renal insufficiency with clearance <30 ml / min / 1.73 m², probability of convulsions during the higher examination in patients with epilepsy or brain injury, pregnancy, breastfeeding;
* Contraindication to MRI: ferromagnetic material (including pacemaker, implantable defibrillators, cardiac valve prostheses, cochlear implants, neurostimulators, implanted automated injection equipment, intraocular metallic foreign bodies, neurosurgical and vascular clips);
* Carotid occlusion;
* ipsilateral intracranial stenosis;
* Risk of pregnancy or proven pregnancy on interrogation data. Breastfeeding;
* Patient under guardianship, under curatorship or safeguard of justice;
* inability to express consent;
* uncontrolled cardiological or neurological diseases;
* Impossibility of being followed for medical, social, geographical or psychological reasons throughout the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
decreased intensity of IPH levels measured by MRI | Day 0
  Image quality will be assessed from 1 to 5 (grade 1, low Signal-to-Noise Ratio (SNR) limits use, arterial wall and vessel margins are unidentifiable; grade 2, marginal SNR, arterial wall is visible, but the substructure, lumen, and outer boundaries are indistinct; grade 3, marginal SNR, wall structures are identifiable, but lumen and outer boundaries are partially obscured; grade 4, high SNR with minimal artifacts, vessel wall, lumen, and adventitial margins are well defined; and grade 5, high SNR without artifacts, wall architecture depicted in detail, lumen and adventitial boundary are clearly defined) . If the quality of the image is sufficient (≥ 3), IPH levels will be semi-quantified on a scale from 0 to 3 (0: No IPH, 1: light IPH, 2 moderate IPH, strong IPH). Images will be assessed blindly and independently by clinical experts of carotid plaque imaging.
decreased intensity of IPH levels measured by MRI | Month 6
  Image quality will be assessed from 1 to 5 (grade 1, low Signal-to-Noise Ratio (SNR) limits use, arterial wall and vessel margins are unidentifiable; grade 2, marginal SNR, arterial wall is visible, but the substructure, lumen, and outer boundaries are indistinct; grade 3, marginal SNR, wall structures are identifiable, but lumen and outer boundaries are partially obscured; grade 4, high SNR with minimal artifacts, vessel wall, lumen, and adventitial margins are well defined; and grade 5, high SNR without artifacts, wall architecture depicted in detail, lumen and adventitial boundary are clearly defined) . If the quality of the image is sufficient (≥ 3), IPH levels will be semi-quantified on a scale from 0 to 3 (0: No IPH, 1: light IPH, 2 moderate IPH, strong IPH). Images will be assessed blindly and independently by clinical experts of carotid plaque imaging.

SECONDARY OUTCOMES:
Evaluation of intermediate monocyte phenotype (cluster of differentiation 14 (CD14)++ /cluster of differentiation 16 (CD16)+) | Day 0
  monocytes will be extracted from blood sample, marked with specific antibodies (anti CD14/16) and intermediate phenotypes (in %) will be measured by flow cytometry
Evaluation of intermediate monocyte phenotype (cluster of differentiation 14 (CD14)++ /cluster of differentiation 16 (CD16)+) | Month 6
  monocytes will be extracted from blood sample, marked with specific antibodies (anti CD14/16) and intermediate phenotypes (in %) will be measured by flow cytometry
Evaluation of classical monocyte phenotype (cluster of differentiation 14 (CD14)++ /cluster of differentiation 16 (CD16)-) | Day 0
  monocytes will be extracted from blood sample, marked with specific antibodies (anti CD14/16) and classical phenotypes (in %) will be measured by flow cytometry
Evaluation of classical monocyte phenotype (cluster of differentiation 14 (CD14)++ /cluster of differentiation 16 (CD16)-) | Month 6
  monocytes will be extracted from blood sample, marked with specific antibodies (anti CD14/16) and classical phenotypes (in %) will be measured by flow cytometry
Evaluation of non-classical monocyte phenotype (cluster of differentiation 14 (CD14)+ /cluster of differentiation 16 (CD16)++) | Day 0
  monocytes will be extracted from blood sample, marked with specific antibodies (anti CD14/16) and non-classical phenotypes (in %) will be measured by flow cytometry
Evaluation of non-classical monocyte phenotype (cluster of differentiation 14 (CD14)+ /cluster of differentiation 16 (CD16)++) | Month 6
  monocytes will be extracted from blood sample, marked with specific antibodies (anti CD14/16) and non-classical phenotypes (in %) will be measured by flow cytometry
Assessment of red blood cell aggregation | Day 0
  Red blood cell aggregation (in %)will be measured by ektacytometry
Assessment of red blood cell aggregation | Month 6
  Red blood cell aggregation (in %) will be measured by ektacytometry
in vitro clotting formation time | Day 0
  In vitro clotting formation time (in minutes) will be measured on whole blood by rotational thromboelastometry
in vitro clotting formation time | Month 6
  In vitro clotting formation time (in minutes) will be measured on whole blood by rotational thromboelastometry
Measurement of in vitro clot lysis index | Day 0
  In vitro clot lysis index (in millimeter) will be measured on whole blood by rotational thromboelastometry
Measurement of in vitro clot lysis index | Month 6
  In vitro clot lysis index (in millimeter) will be measured on whole blood by rotational thromboelastometry
Measurement of in vitro clot firmness | Day 0
  In vitro clot firmness (in millimeter) will be measured on whole blood by rotational thromboelastometry
Measurement of in vitro clot firmness | Month 6
  In vitro clot firmness (in millimeter) will be measured on whole blood by rotational thromboelastometry
Assessment of plasma lipid oxidation | Day 0
  Plasma protein oxidation (advanced oxidation proteins products) measured by by spectrophotometry (in micromole/liter (µmol/L))
Assessment of plasma lipid oxidation | Month 6
  Plasma protein oxidation (advanced oxidation proteins products) measured by by spectrophotometry (in micromole/liter (µmol/L))
Assessment of plasma protein oxidation | Day 0
  Plasma protein oxidation (advanced oxidation proteins products) measured by by spectrophotometry (in micromole/liter (µmol/L))
Assessment of plasma protein oxidation | Month 6
  Plasma protein oxidation (advanced oxidation proteins products) measured by by spectrophotometry (in micromole/liter (µmol/L))
Assessment of plasma protein nitration | Day 0
  Plasma protein nitration (nitrotyrosine) measured by the enzyme-linked immunosorbent assay (ELISA) in micromole/liter (µmol/L).
Assessment of plasma protein nitration | Month 6
  Plasma protein nitration (nitrotyrosine) measured by the enzyme-linked immunosorbent assay (ELISA) in micromole/liter (µmol/L).
Assessment of plasma inflammatory markers | Day 0
  Plasma inflammatory markers will be measured by multiplex assay in micromole/liter (µmol/L).
Assessment of plasma inflammatory markers | Month 6
  Plasma inflammatory markers will be measured by multiplex assay in micromole/liter (µmol/L).
Assessment of plasma enzymes activity | Day 0
  Plasma antioxidant enzymes activity will be measured by enzymology (in micromole/liter/minute (µmol/L/min))
Assessment of plasma enzymes activity | Month 6
  Plasma antioxidant enzymes activity will be measured by enzymology (in micromole/liter/minute (µmol/L/min))
number of steps per day | during 2 weeks after Day 0
  the daily number of steps (in number of step per day) will be measured using a connected wrist activity tracker
number of steps per day | during 2 weeks after Month 6
  the daily number of steps (in number of step per day) will be measured using a connected wrist activity tracker
distance of the 6 minutes walking test | Day 0
  The distance at the 6 minutes walking test (in meters) will be evaluated on the 30meters flat round-trip
distance of the 6 minutes walking test | Month 6
  The distance at the 6 minutes walking test (in meters) will be evaluated on the 30meters flat round-trip
quadriceps maximal isometric strength | Day 0
  The quadriceps maximal isometric strength (in Newton) will be evaluated in sitting position using dynamometer
quadriceps maximal isometric strength | Month 6
  The quadriceps maximal isometric strength (in Newton) will be evaluated in sitting position using dynamometer
Determination of the level of physical activity | Day 0
  the level physical activity will be evaluated by the global physical activity questionnaire (in Metabolic Equivalent of Task/minutes per week (MET/min.week)).
Determination of the level of physical activity | Month 6
  the level physical activity will be evaluated by the global physical activity questionnaire (in Metabolic Equivalent of Task/minutes per week (MET/min.week)).
Determination of the sedentary time | Day 0
  Sedentary time will be evaluated by the sedentary behaviour questionnaire evaluating the total daily sitting and lying down time (in minute/day) during awaking time.
Determination of the sedentary time | Month 6
  Sedentary time will be evaluated by the sedentary behaviour questionnaire evaluating the total daily sitting and lying down time (in minute/day) during awaking time.
descriptive health state score | Day 0
  Health state score will be assessed using descriptive system of the EQ-5D-5L (five-level version of the EuroQol five-dimensional) questionnaire.
  Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The subjects self-rate their level of severity for each dimension using a five-level (EQ-5D-5L) scale (scored from 1 to 5, 1 indicating no problem and 5 indicating extreme problem).
  The health rate score correspond to the addition of each dimension score and is from 5 to 25. The lower the score, the better the health state.
descriptive health state score | Month 6
  Health state score will be assessed using descriptive system of the EQ-5D-5L (five-level version of the EuroQol five-dimensional) questionnaire.
  Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The subjects self-rate their level of severity for each dimension using a five-level (EQ-5D-5L) scale (scored from 1 to 5, 1 indicating no problem and 5 indicating extreme problem).
  The health rate score correspond to the addition of each dimension score and is from 5 to 25. The lower the score, the better the health state.
self-evaluated overall health status | Day 0
  Overall health status will be assessed using the evaluation part of the EQ-5D-5L (five-level version of the EuroQol five-dimensional) questionnaire.
  The subject's self- evaluate their overall health status using the visual analogue scale (EQ-VAS).
  The raw score is from 0 to 100. The higher the score, the better the perceived overall health status
self-evaluated overall health status | Month 6
  Overall health status will be assessed using the evaluation part of the EQ-5D-5L (five-level version of the EuroQol five-dimensional) questionnaire.
  The subject's self- evaluate their overall health status using the visual analogue scale (EQ-VAS).
  The raw score is from 0 to 100. The higher the score, the better the perceived overall health status
body mass index | Day 0
  Body mass index (in kilogram/metre² (kg/m²)) will be calculated with the measurement of body weight (in kilogram) and height (in meter)
body mass index | Month 6
  Body mass index (in kilogram/metre² (kg/m²)) will be calculated with the measurement of body weight (in kilogram) and height (in meter)
number of comorbidities | Day 0
  Number of comorbidities (Diabetes, hypertension, obesity and , poly-atheroma) will be determined
number of comorbidities | Month 6
  Number of comorbidities (Diabetes, hypertension, obesity and , poly-atheroma) will be determined

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France

REFERENCES:
- [Result] Mura M, Rivoire E, Dehina-Khenniche L, Weiss-Gayet M, Chazaud B, Faes C, Connes P, Long A, Rytz CL, Mury P, Delrieu L, Gouraud E, Bordet M, Della Schiava N, Lermusiaux P, Arsicot M, Millon A, Pialoux V. Effectiveness of an individualized home-based physical activity program in surgery-free non-endarterectomized asymptomatic stroke patients: a study protocol for the PACAPh interventional randomized trial. Trials. 2022 Feb 14;23(1):145. doi: 10.1186/s13063-022-06061-x. PMID 35164816
- [Result] Mura M, Rivoire E, Dehina-Khenniche L, Jazzar G, Schlatter S, Della-Schiava N, Arsicot M, Fayad ZA, Lermusiaux P, Long A, Douek P, Chirico EN, Thomas A, Pialoux V, Millon A. Influence of a six-month home-based individualized physical activity intervention on carotid plaque instability measured by magnetic resonance imaging: a randomized controlled clinical trial. EClinicalMedicine. 2025 Apr 22;83:103158. doi: 10.1016/j.eclinm.2025.103158. eCollection 2025 May. PMID 40548131